CLINICAL TRIAL: NCT06722404
Title: Effect of Synbiotics on Hematological Indices of Malnourished Children
Brief Title: Synbiotics for the Management of Malnutrition (Children)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BeSt 44/ 17; PIN No. 085-14090-AV5-176 (Other Grant/Funding Number: Higher Education Commission (HEC), Pakistan)
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition | interventions — Synbiotics

STUDY DESIGN:
Intervention Model Description: All children were initially fed F-75 (75 kcal/ 100mL) therapeutic milk (Phase I) and then progressed to F-100 (100 kcal/ 100mL) (Phase II) and Plumpy'nuts (F-100 in spread form with iron fortification) (Phase III) with follow-up for 48 days. Synbiotics treatments were given from the onset of F-75 till the child progressed.The control group received standard therapeutic foods (F-75, F-100 and Plumpy'nuts), whereas the intervention group received therapeutic foods plus synbiotics containing Oligomate that was fortified in F75 at the rate of 7.5 g/L containing 4.1 g/L GOS for 1 g/100 kcal dose and at the rate of 11.5 g/L containing 6.1 g/L GOS for 1.5 g/100 kcal dose while in F100 and Plumpy'nuts it was fortified at the rate of 10 g/L containing 5.5 g/L GOS for 1 g/100 kcal dose
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard therapeutic food group (Active Comparator): The control group received standard therapeutic foods (F-75, F-100 and Plumpy'nuts)
  Interventions: Dietary Supplement: Standard therapeutic foods
- therapeutic foods plus synbiotics group (Experimental): the intervention group received therapeutic foods plus synbiotics containing Oligomate that was fortified in F75 at the rate of 7.5 g/L containing 4.1 g/L GOS for 1 g/100 kcal dose and at the rate of 11.5 g/L containing 6.1 g/L GOS for 1.5 g/100 kcal dose while in F100 and Plumpy'nuts it was fortified at the rate of 10 g/L containing 5.5 g/L GOS for 1 g/100 kcal dose and at the rate of 15 g/L containing 8.25 g/L GOS for 1.5 g/100 kcal dose and Resiton (Lactobacillus paracasei sbsp. paracasei) 3 billion cfu/day and 6 billion cfu/day that were mixed in different combinations.
  Interventions: Combination Product: Therapeutic foods plus Synbiotics

INTERVENTIONS:
Dietary Supplement: Standard therapeutic foods — All children were initially fed F-75 (75 kcal/ 100mL) therapeutic milk (Phase I) and then progressed to F-100 (100 kcal/ 100mL) (Phase II) and Plumpy'nuts (F-100 in spread form with iron fortification) (Phase III) with follow-up for 48 days
  Arms: standard therapeutic food group
Combination Product: Therapeutic foods plus Synbiotics — the intervention group received therapeutic foods plus synbiotics containing Oligomate that was fortified in F75 at the rate of 7.5 g/L containing 4.1 g/L GOS for 1 g/100 kcal dose and at the rate of 11.5 g/L containing 6.1 g/L GOS for 1.5 g/100 kcal dose while in F100 and Plumpy'nuts it was fortified at the rate of 10 g/L containing 5.5 g/L GOS for 1 g/100 kcal dose and at the rate of 15 g/L containing 8.25 g/L GOS for 1.5 g/100 kcal dose and Resiton (Lactobacillus paracasei sbsp. paracasei) 3 billion cfu/day and 6 billion cfu/day that were mixed in different combinations.
  Arms: therapeutic foods plus synbiotics group

SUMMARY:
In this study, dose related effect of synbiotics on the blood indices of severely acute malnourished (SAM) children (6-59 months) was carried out in hospitalized setting. Fifty SAM children were enrolled in a double-blind, randomized design.

DETAILED DESCRIPTION:
The study was done at Nutrition Rehabilitation Unit (NRU), Department of Social & Preventive Pediatrics, Mayo Hospital, Lahore, Pakistan, a Tertiary Care large urban teaching and referral hospital and was approved by human ethics Institutional Review Board (IRB) .Galacto-oligosaccharides (Oligomate) as prebiotics were procured from Yakult Pharmaceutical Industry, Japan and Resiton (lactobacillus paracasei subsp. paracasei) as probiotics were procured from MakNsons Pharmaceutical Industry, Italy. In the present study we enrolled 50 severely acute malnourished (SAM) in patients of 6-59 months of age while follow-up treatment was given at the out-patient department. We define SAM as weight-for height of less than 70% of the median, nutritional edema (Kwashiorkor), or both, mid-upper arm circumference (MUAC) of less than 11.5cm. Anthropometry protocols were followed by research standards

ELIGIBILITY:
Inclusion Criteria:

* In the present study we enrolled 50 severely acute malnourished (SAM) patients of 6-59 months of age while follow-up treatment was given at the out-patient department.

  * Patients having weight-for-height of less than 70% of the median, nutritional edema (Kwashiorkor), or both,
  * mid-upper arm circumference (MUAC) of less than 11.5cm

Exclusion Criteria:

* Participant taking other supplements or enrolled in other studies

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Weight | 48 days
  weight change observed in patients
Number of Stools | 48 days
  Number of stools per day

SECONDARY OUTCOMES:
Complete blood count (CBC) | 48 days
  For hematological and biochemical screening 5 mL venous blood was taken after 12 h fasting in vacutainers tubes containing ethylenediamine tetra-acetic acid (EDTA). Complete blood count (CBC) was carried out using haemocytometer
Serum albumin levels | 48 days
  The assay is based on the selective interaction between BCG and albumin forming a chromophore that can be detected at 620 nm using spectrophotometer. The signal is directly proportional to the amount of albumin present in the serum. BCG does not react with other abundant plasma proteins like IgG
serum electrolytes | 48 days
  Serum electrolytes such as Na and K were analyzed by electrolyte analyzer (Biolyte 2000; BioCare Corporation, Taiwan). Briefly, 10 mL blood was obtained from each subject and then blood samples were allowed to stand for 1 h to clot. Thereafter, blood samples were centrifuged at 300 rpm, 15 min at room temperature. The supernatant was then separated from the settled bottom blood cells
ESR determination | 48 days
  anti-coagulated blood was allowed to stand in a narrow vertical glass tube, undisturbed for a period of time, the RBCs under the influence of gravity settled out from the plasma. The rate at which they settled was measured as the number of millimeters of clear plasma present at the top of the column after one hour (mm/h).
SGPT/ ALT | 48 days
  ALT is an important indicator of liver disease. The series of reactions involved in the assay system is as follows; L-Alanine + 2- oxoglutarate → Pyruvate + L-Glutamate; Pyruvate + NADH → Lactate+ NAD. Then this rate of Nicotinamide adenine dinucleotide (NADH) consumption is determined photo metrically that is proportional to ALT activity in the sample.
SGOT/ AST | 48 days
  The AST is the cellular enzyme, is found in highest concentration in heart muscle, the cells of the liver and the cells of the skeletal muscle. The rate of decrease in concentration of NADH, measured photometrically at 340 nm is proportional to the catalytic concentration of AST present in the sample.
Alkaline Phosphatase | 48 days
  For the determination of alkaline phosphatase, the following protocol was adopted . Alkaline phosphatase release phenol from para nitrophenylphosphate, the phenol in alkaline medium gives yellow color which can be estimated with spectrophotometer at 405 nm. The reagents required for this experiment are R1=diethanolamine (pH 9.8, 1.2 mol/L), magnesium chloride (0.6 mmol/L); R2=p-nitrophenylphosphate (50 mmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Habib Ur Rehman, Principal Investigator — University of Veterinary and Animal Sciences,Lahore
Locations (1):
- Nutrition Rehabilitation Unit (NRU), Department of Social & Preventive Pediatrics, Mayo Hospital,, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
study data will be published in research journal without personal identity

REFERENCES:
- [Background] Basu S, Chatterjee M, Ganguly S, Chandra PK. Effect of Lactobacillus rhamnosus GG in persistent diarrhea in Indian children: a randomized controlled trial. J Clin Gastroenterol. 2007 Sep;41(8):756-60. doi: 10.1097/01.mcg.0000248009.47526.ea. PMID 17700424